CLINICAL TRIAL: NCT04232579
Title: Diagnosis of Asthma, COPD and ACO in Vietnamese Context, Proposal of a Therapeutic Strategy Compatible With the Guidelines and Development of Predictive Biomarkers of the Response to Treatment
Brief Title: Development of Predictive Biomarkers for the Diagnosis and Treatment of Asthma and COPD in Vietnam.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Olivier Michel (Other)
Responsible Party: Sponsor-Investigator, Olivier Michel, Head of Immuno-allergology department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: ACORD
Record Dates: First submitted 2019-12-05; First posted 2020-01-18 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Respiratory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic obstructive respiratory disease: The out-patient population with chronic obstructive respiratory disease consulted at Nguyen Tri Phuong Hospital, Ho Chi Minh city, Vietnam.
  Interventions: Other: Therapeutic strategy

INTERVENTIONS:
Other: Therapeutic strategy — Therapeutic strategy compatible with the guidelines and development of predictive biomarkers of the response to treatment.

SUMMARY:
According to World Health Organization (WHO), non-communicable diseases account for 70% of global mortality. Chronic Respiratory Disease (CRD) affects more than one billion people and is the third leading cause of annual death of five million people after cardiovascular disease and cancer. Asthma and chronic obstructive pulmonary disease (COPD) are the two most common diseases of CRD and are part of obstructive airway disease (OAD).

Asthma and COPD are distinguished by the clinical manifestations and therapeutic strategy according to Global Initiative for Asthma (GINA) and Global Initiative for Chronic Obstructive Lung Disease (GOLD). However, in Vietnam, most patients with OAD are treated with an inhaled corticosteroid (ICS) combined with a long-lasting bronchodilator because the specific diagnosis is not always possible.

In addition, a significant proportion of patients have clinical features of both asthma and COPD that is defined as the asthma COPD overlap (ACO). The definition of ACO remains controversial because it is not a distinct disease in which their specific treatment is still under debate that ICS is being generally proposed.

It is understood that most OAD in Vietnam is treated with ICS. However, it is now accepted that in COPD (or COPD-like ACO) patients receiving this treatment may promote respiratory infections and even tuberculosis in endemic countries including Vietnam.

Few data on the relative prevalence of asthma, COPD, and ACO are available in Vietnam. A recent study in Vietnam proposed defining asthma, COPD and ACO based on symptoms, ventilatory obstruction and bronchodilator (BD) reversibility, cumulative smoking, and age. Mites sensitization and exposure to biomass fume were then evaluated in patients having ACO. By doing so, COPD patients are smoking (≥ 10 pack-years) and have irreversible bronchial obstruction. Asthmatics are those with completely reversible bronchial obstruction OR non-smoking patients (<10 pack-years) and partially reversible obstructive. The other OAD patients were classified as having "ACO". Based on these definitions, the prevalence of COPD, asthma and ACO was 40%, 18% and 42%, respectively. Then ACO was defined as "from COPD, or ACO-COPD" in case of biomass exposure and negative mite skin tests, the others being ACO "from asthma or ACO-asthma".

Currently, several biomarkers have been evaluated in the differential diagnosis and prognosis of OAD. The concentration of immunoglobulin E (IgE), the number of eosinophils in blood and sputum, nitric oxide (NO) in exhaled air, and recently periostin have been associated with asthma. On the other hand, biomarkers of systemic inflammation (C-reactive protein (CRP), fibrinogen, TNFα, IL-6 and IL-8) have also been investigated in COPD. Few data are available on the ACO biomarkers.

In this study, the investigators will define the different phenotypes of chronic OAD (asthma, ACO-asthma, ACO-COPD and COPD) taking into account the reversibility of bronchial obstruction, cumulative smoking, biomass fume exposure and immediate sensitization to mites. Blood biomarkers and exhaled NO will be measured and analyzed in each phenotype.

The treatment of COPD, asthma, ACO-COPD, and ACO-asthma based on the GINA and GOLD recommendations will be compared to the current practice in Vietnam: use of ICS with or without long-acting beta-agonists (LABA).

Specific biomarkers will also be evaluated as predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* Signed informed consent
* Out-patients at Nguyen Tri Phuong Hospital
* One or several symptoms suggesting chronic respiratory disease (cough, chest tightness, wheezing, dyspnea or sputum), lasting 3 months or more.
* Lung function abnormality (Forced Expiratory Volume in 1 Second /Forced Vital Capacity < Lower Limit of Normal)
* Patients are able to stop anti-histamine 5 days before evaluation
* Patients are able to stop bronchodilator treatment before performing lung function test according to standard practice (immediate release theophylline: 24 hours, long acting β2-agonist: 12 hours, short acting β2-agonist: 6 hours and short acting anticholinergic: 8 hours).

Exclusion Criteria:

* Presence of one or more chronic diseases: HIV infection, active tuberculosis, heart failure, cancers, auto-immune diseases, systemic diseases, low BMI (<18.5) or mental health disorders.
* Treatment with non-selective beta-blockers
* Severe exacerbation during the last month
* Corticosteroid-dependent patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The out-patient population with chronic obstructive respiratory disease consulted at Nguyen Tri Phuong Hospital, Ho Chi Minh city, Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Relative prevalence of the different chronic obstructive respiratory disease phenotypes. | 12 months after the start of the study
  The relative prevalence will be measured by the percentage of each phenotype of chronic respiratory diseases, according to lung function test, cumulative smoking, mite sensitization on prick tests and biomass fume exposure.
Asthma Control Test | 26 months after start of study
  Questionnaire: 5 questions scored according to a 5 point Likert Scale. Total inferior to 15: uncontrolled asthma. Between 15 and 19: partially controled asthma. From 20 to 25: controled asthma.
COPD Assessment Test | 26 months after start of study
  Questionnaire that contains eight questions covering domains relating to the impact of COPD symptoms. Scores of 0-10, 11-20, 21-30, 31-40 represent mild, moderate, severe or very severe clinical impact.
Asthma Quality of Life Questionnaire | 26 months after start of study
  A disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease. The scoring follows a 7-point Likert scale (7 = not impaired at all - 1 = severely impaired).
Number of exacerbations | 26 months after start of study
  Number of exacerbations
Spirometry results | 26 months after start of study
  Spirometry is the most common of the pulmonary function tests. Spirometry generates pneumotachographs, which are charts that plot the volume and flow of air coming in and out of the lungs from one inhalation and one exhalation.

SECONDARY OUTCOMES:
White blood cells count (WBC) | 12 months after the start of the study
  White blood cells count
White blood cells count (WBC) | 26 months after the start of the study
  White blood cells count
C-reactive protein (CRP) | 12 months after the start of the study
  C-reactive protein (CRP) level in blood
C-reactive protein (CRP) | 26 months after the start of the study
  C-reactive protein (CRP) level in blood
Erythrocyte sedimentation rate (ESR) | 12 months after the start of the study
  Erythrocyte sedimentation rate in blood
Erythrocyte sedimentation rate (ESR) | 26 months after the start of the study
  Erythrocyte sedimentation rate in blood
IgE concentration | 12 months after the start of the study
  Total IgE concentration in blood
IgE concentration | 26 months after the start of the study
  Total IgE concentration in blood
α1-antitrypsin (A1A) concentration | 12 months after the start of the study
  α1-antitrypsin (A1A) concentration in blood
α1-antitrypsin (A1A) concentration | 26 months after the start of the study
  α1-antitrypsin (A1A) concentration in blood
Fractional exhaled nitric oxide (FENO) | 12 months after the start of the study
  Fractional exhaled nitric oxide
Fractional exhaled nitric oxide (FENO) | 26 months after the start of the study
  Fractional exhaled nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michel, Study Director — CHU Brugmann
Locations (2):
- CHU Brugmann, Brussels, Belgium
- Nguyen Tri Phuong Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee CH, Kim K, Hyun MK, Jang EJ, Lee NR, Yim JJ. Use of inhaled corticosteroids and the risk of tuberculosis. Thorax. 2013 Dec;68(12):1105-13. doi: 10.1136/thoraxjnl-2012-203175. Epub 2013 Jun 8. PMID 23749841
- [Background] Chu HT, Godin I, Phuong NT, Nguyen LH, Hiep TTM, Michel O. Allergen sensitisation among chronic respiratory diseases in urban and rural areas of the south of Viet Nam. Int J Tuberc Lung Dis. 2018 Feb 1;22(2):221-229. doi: 10.5588/ijtld.17.0069. PMID 29506620
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675